CLINICAL TRIAL: NCT06475339
Title: Predicting Responses to Exhausting, Prolonged, And Repeated Exercise Demands (PREPARED) for Heat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Riana Pryor, Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007981; CDMRP-BA230031 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-06-14; First posted 2024-06-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hyperthermia; Fatigue; Heat
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 30/30 work/rest cycle first (Active Comparator): Participants will first complete the 30/30 work/rest cycle, and then complete the other three conditions in a randomized fashion
  Interventions: Other: 30/30 work/rest cycle; Other: 30/20 work/rest cycle; Other: 40/30 work/rest cycle; Other: 20/12 work/rest cycle
- 30/20 work/rest cycle first (Experimental): Participants will first complete the 30/20 work/rest cycle, and then complete the other three conditions in a randomized fashion
  Interventions: Other: 30/30 work/rest cycle; Other: 30/20 work/rest cycle; Other: 40/30 work/rest cycle; Other: 20/12 work/rest cycle
- 40/30 work/rest cycle first (Experimental): Participants will first complete the 40/30 work/rest cycle, and then complete the other three conditions in a randomized fashion
  Interventions: Other: 30/30 work/rest cycle; Other: 30/20 work/rest cycle; Other: 40/30 work/rest cycle; Other: 20/12 work/rest cycle
- 20/12 work/rest cycle first (Experimental): Participants will first complete the 20/12 work/rest cycle, and then complete the other three conditions in a randomized fashion
  Interventions: Other: 30/30 work/rest cycle; Other: 30/20 work/rest cycle; Other: 40/30 work/rest cycle; Other: 20/12 work/rest cycle

INTERVENTIONS:
Other: 30/30 work/rest cycle — Participants will walk on a treadmill while wearing a weighted backpack to a work/rest cycle of 30 minutes of work followed by 30 minutes of rest.
Other: 30/20 work/rest cycle — Participants will walk on a treadmill while wearing a weighted backpack to a work/rest cycle of 30 minutes of work followed by 20 minutes of rest.
Other: 40/30 work/rest cycle — Participants will walk on a treadmill while wearing a weighted backpack to a work/rest cycle of 40 minutes of work followed by 30 minutes of rest.
Other: 20/12 work/rest cycle — Participants will walk on a treadmill while wearing a weighted backpack to a work/rest cycle of 20 minutes of work followed by 12 minutes of rest.

SUMMARY:
The overall goal of this project is to identify a work/rest cycle that allows for faster mission completion needed in emergency situations, compared to current Army heat guidance, while mitigating heat strain and neuromuscular fatigue. This project will determine the trade-off between faster mission completion and risk of heat strain and physical performance decrements. Completion of this project will allow military leaders to make informed decisions by understanding the impact of their choices on the magnitude of physical performance decrements and expected heat casualties, setting up hot weather missions for success.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Physically active

Exclusion Criteria:

* History of cardiovascular, metabolic (such as clinical thyroid disease), respiratory, neural, or renal disease
* Hypertensive (systolic blood pressure > 139 mmHg, diastolic blood pressure > 89 mmHg) or tachycardic (heart rate > 100 bpm) during the screening visit
* Taking medications or supplements known to effect physiologic responses to exercise or thermoregulation (e.g., beta blockers, omega-3 fatty acids, statins, aspirin)
* Tobacco or nicotine use currently or in the past six months
* Musculoskeletal injury expected to impact exercise in the protocol
* A positive pregnancy test at any point in the study
* Study physician discretion based on any other medical condition or medication
* Inability to understand or follow instructions or the protocol
* Gastrointestinal disease or previous surgery prohibiting core temperature capsule use. Participants with a contraindication can opt to insert the pill rectally as a suppository.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Core temperature | 180 minutes of work
  Maximum gastrointestinal temperature reached during the work protocol
Isometric mid-thigh pull strength | 180 minutes of work
  Maximum voluntary contraction strength assessed using a force plate

SECONDARY OUTCOMES:
Metabolic cost | 180 minutes of work
  Collected expired air using a one-way mask will be analyzed using a metabolic cart to calculate metabolic heat production
Heart rate | 180 minutes of work
  Maximum heart rate measured using a telemetry strap throughout the work protocol
Mean skin temperature | 180 minutes of work
  Maximum skin temperature measured using buttons at four skin sites
Vastus lateralis electromyography | 180 minutes of work
  Wireless electromyography electrodes placed lengthwise over the vastus lateralis muscle belly

CONTACTS AND LOCATIONS:
Overall Officials: Riana R Pryor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Center for Research and Education in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be shared via publications and/or presentations. De-identified data may be shared and reviewed by the Department of Defense and as part of our Cooperative Research & Development Agreement with the United States Army Research Institute of Environmental Medicine.